CLINICAL TRIAL: NCT04899908
Title: A Double-blind, Phase II Randomized Study of Brain-directed Stereotactic Radiation With or Without AGuIX Gadolinium-based Nanoparticles in the Management of Brain Metastases at Higher Risk of Local Recurrence With Radiation Alone
Brief Title: Stereotactic Brain-directed Radiation With or Without Aguix Gadolinium-Based Nanoparticles in Brain Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: NH TherAguix SAS (Other)
Responsible Party: Principal Investigator, Ayal Aizer, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20-240
Record Dates: First submitted 2021-04-30; First posted 2021-05-25 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Brain Cancer; Brain Metastases; Melanoma; Lung Cancer; Breast Cancer; HER2-positive Breast Cancer; Colorectal Cancer; Gastrointestinal Cancer; SRS; SRT; Whole Brain Radiation; Stereotactic Radiation; AGuIX; Nanoparticle; Cystic; Brain Tumor
Keywords: Brain Cancer; Brain Metastases; Melanoma; Lung Cancer; Breast Cancer; HER2-positive Breast Cancer; Colorectal Cancer; Gastrointestinal Cancer; SRS; SRT; Whole brain radiation; Stereotactic Radiation; AGuIX; Nanoparticle; Cystic; Brain Tumor
MeSH Terms: conditions — Brain Neoplasms; Melanoma; Lung Neoplasms; Breast Neoplasms; Colorectal Neoplasms; Gastrointestinal Neoplasms | interventions — Radiosurgery; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Stereotactic Radiation plus AGuIX gadolinium-based nanoparticles (Experimental): Randomly assigned participants will receive:
  * AGuIX gadolinium-based nanoparticles 3-5 days before radiation is initiated
  * AGuIX gadolinium-based up to 2x during radiation, depending on standard of care radiation treatment.
    * If standard of care radiation treatment involves only one day of radiation, participant will receive AGuIX gadolinium-based nanoparticles on the day of radiation.
    * If standard of care radiation treatment involves 5 or 6 days of radiation, participant will receive AGuIX gadolinium-based nanoparticles two-times (2x) in total, on the first and third day of radiation.
  Interventions: Radiation: Stereotactic Radiation; Drug: AGuIX gadolinium-based nanoparticles
- Stereotactic Radiation plus placebo (Experimental): Randomly assigned participants will receive:
  * Placebo 3-5 days before radiation is initiated
  * Placebo up to 2x during radiation, depending on standard of care radiation treatment.
    * If standard of care radiation treatment involves only one day of radiation participant will receive Placebo on the day of radiation.
    * If standard of care radiation treatment involves 5 or 6 days of radiation participant will receive Placebo two-times (2x) in total, on the first and third day of radiation.
  Interventions: Radiation: Stereotactic Radiation; Other: Placebo

INTERVENTIONS:
Radiation: Stereotactic Radiation — Focused radiation beams to treat tumors
  Other Names: Stereotactic Radiotherapy
Drug: AGuIX gadolinium-based nanoparticles — Intravenous injection
  Arms: Stereotactic Radiation plus AGuIX gadolinium-based nanoparticles
Other: Placebo — Intravenous infusion
  Other Names: Saline
  Arms: Stereotactic Radiation plus placebo

SUMMARY:
The purpose of this study is to determine whether AGuIX (Activation and Guidance of Irradiation by X-ray) gadolinium-based nanoparticles make radiation work more effectively in the treatment of patients with brain metastases that are more difficult to control with stereotactic radiation alone.

DETAILED DESCRIPTION:
This research study is a double-blind, randomized phase II clinical trial of brain-directed stereotactic radiation with or without AGuIX (Activation and Guidance of Irradiation by X-ray) gadolinium-based nanoparticles in the management of brain metastases at higher-risk of local recurrence with radiation alone.

The study agent (AGuIX gadolinium-based nanoparticles) has two main parts. The first is gadolinium, also known as "contrast," which is typically injected into a vein during a MRI scan. The second part is a nanoparticle (linked to the gadolinium) that may make focused radiation work more effectively. The AGuIX gadolinium-based nanoparticles are deposited within the brain metastases via the bloodstream and then the brain metastases are radiated.

The U.S. Food and Drug Administration (FDA) has not approved AGuIX gadolinium-based nanoparticles as a treatment for any disease. AGuIX gadolinium-based nanoparticles have been tested in other studies for safety and efficacy in patients with brain metastases who are also receiving radiation.

This study seeks to determine whether AGuIX gadolinium-based nanoparticles improve outcomes relative to placebo.Participants will be "randomized" into one of the study groups:

* Group A: Radiation plus AGuIX gadolinium-based nanoparticles
* Group B: Radiation plus placebo

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

NH TherAguix, the manufacturer of the AGuIX gadolinium-based nanoparticles, is supporting this research study by providing the AGuIX gadolinium-based nanoparticles that will be evaluated in this study.

NH TherAguix is also covering the cost of the study.

It is expected that about 134 people will take part in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a biopsy proven solid malignancy and at least one intracranial measurable lesion spanning ≥5mm in maximal unidimensional size and radiographically consistent with or pathologically proven to be a brain metastasis AND meet one of the following additional criteria regarding the primary site or nature of the intracranial disease:

  * Melanoma with intracranial growth consistent with tumor progression despite immunotherapy
  * Gastrointestinal primary
  * HER2 positive breast cancer (subtype assessed using most representative tissue available in opinion of enrolling clinician and/or study PI)
  * Cystic metastases
  * Metastases ≥2cm in maximal unidimensional size
  * Locally recurrent metastases after prior stereotactic radiation
  * Locally recurrent metastases after prior whole brain radiation *Patients with metastases from melanoma, GI primaries, or HER2+ breast cancer, as well as those with cystic metastases or metastases ≥2cm in maximal unidimensional size, who have local recurrences after prior brain-directed radiation can only be treated in the strata permitting prior radiation (last two strata above)
* Age ≥18 years at diagnosis of brain metastases
* Estimated glomerular filtration rate of ≥ 60 mL/min/1.73m2
* Karnofsky performance status of at least 70 (i.e. at minimum, "cares for self" but "unable to carry on normal activity or do active work")
* Estimated survival based on extracranial disease of at least 3 months in the opinion of the enrolling clinician and/or study PI
* Ability to understand and the willingness to sign a written informed consent document
* The effects of AGuIX on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception prior to study entry and for the duration of the therapeutic component of study participation

Exclusion Criteria:

* Participants who cannot undergo a brain MRI
* Participants who cannot receive gadolinium
* Participants with widespread, definitive leptomeningeal disease
* Patients requiring radiation to either >10 targets (if naïve to whole brain radiation) or >20 targets (if whole brain radiation has been given previously) per the discretion of the treating clinician and/or study PI
* Pregnant women are excluded from this study because of the potential deleterious effects of gadolinium on the developing fetus. Because there is an unknown but potential risk for adverse events in nursing infants, women who are breastfeeding are not eligible for this study
* In cohorts who have received prior brain-directed radiation, patients are not eligible for this study if they have active (at the time of protocol screening) brain metastases that require radiation that are in or within 1.0cm of the brainstem, eyes, optic nerves, or optic chiasm if the juxtaposed organ at risk (i.e. brainstem, eyes, optic nerves, or optic chiasm) has previously received either >6.0 Gy in a single fraction or, if prior radiation was fractionated, a cumulative dose in 2.0 Gy equivalents, using an alpha/beta ratio of 2, of >40.0 Gy. In addition, all patients who have had prior brain-directed radiation, regardless of technique/dose/fractionation, are not eligible for the study until written approval is provided by the study/site PI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Local Recurrence | From enrollment to 6 months
  Assessed with Response Assessment in Neuro-Oncology (RANO) - Brain Metastasis Guidelines Time to local failure on a per metastasis basis will be performed using the log-rank test.

SECONDARY OUTCOMES:
Overall Survival (OS) | Time from enrollment to 12 months
  Assessed with log-rank test
Progression-Free Survival (PFS) | Time from enrollment to 12 months
  Assessed with log-rank test
Time to Progression (TTP) | Time from enrollment to 12 months
  Assessed with log-rank test
Death due to neurologic causes | From enrollment to 12 months
  Assessed with Gray's test
Performance status | From enrollment to 12 months
  Karnofsky performance status, assessed longitudinally (longitudinal regression)
Ability to complete activities of daily living | From enrollment to 12 months
  Questionnaire - EQ-5D, assessed longitudinally (longitudinal regression)
Incidence and time to detection of new brain metastases | From enrollment to 12 months
  Assessed with log-rank test
Incidence and time to detection of radiation necrosis | From enrollment to 12 months
  Assessed with log-rank test
Incidence and time to detection of leptomeningeal disease | From enrollment to 12 months
  Assessed with log-rank test
Incidence and time to detection of progressive intracranial disease | From enrollment to 12 months
  Assessed with log-rank test
Incidence and time to detection of salvage craniotomy | From enrollment to 12 months
  Assessed with log-rank test
Incidence and time to additional radiotherapeutic treatments | From enrollment to 12 months
  Assessed with log-rank test
Incidence and time to the development of seizures | From enrollment to 12 months
  Assessed with log-rank test
Steroid use | From enrollment to 12 months
  Assessed longitudinally (longitudinal regression)
Local recurrence at one year in metastases treated radiotherapeutically | From enrollment to 12 months
  Assessed using RECIST (response evaluation criteria in solid tumors) criteria
Neurocognitive function: verbal learning and memory | From enrollment to 12 months
  Hopkins Verbal Learning Test - Revised (HVLT-R)
Neurocognitive function: visual attention and task switching | From enrollment to 12 months
  Trail Making Test Part A and B (TMT)
Neurocognitive function: verbal fluency | From enrollment to 12 months
  Controlled Word Association Test (COWAT)
Neurocognitive function: cognitive impairment | From enrollment to 12 months
  Mini Mental Status Examination (MMSE)

CONTACTS AND LOCATIONS:
Overall Officials: Ayal Aizer, MD, MHS, Principal Investigator — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Derived] Bennett S, Verry C, Kaza E, Miao X, Dufort S, Boux F, Cremillieux Y, de Beaumont O, Le Duc G, Berbeco R, Sudhyadhom A. Quantifying gadolinium-based nanoparticle uptake distributions in brain metastases via magnetic resonance imaging. Sci Rep. 2024 May 25;14(1):11959. doi: 10.1038/s41598-024-62389-1. PMID 38796495